CLINICAL TRIAL: NCT01704222
Title: Epidemiology of Human Cytomegalovirus Excretion in the Saliva of Children Attending Nursery in France.
Acronym: CrèchMV
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I07040 CrèchMV
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Volunteers
Keywords: Children; nursery; CMV; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Direct DNA amplification, viral isolation and specific antibody measurement in saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Child in nursery: Children older than 3 months and less than 6 years kept in nurseries retained, regardless of the duration of custody of the child in the manger concerned.

SUMMARY:
Direct DNA amplification, viral isolation and specific antibody measurement in saliva from children attending nursery in France Sample collection will be done by the pediatrician the nurse, or one of the authorized investigators of the study.

DETAILED DESCRIPTION:
Salivary collection kit. 3 swab for DNA research, 1 for antibodies research and 1 for virus isolation by cell growth.

ELIGIBILITY:
Inclusion Criteria:

* Children older than 3 months and less than 6 years kept in nurseries retained, regardless of the duration of custody of the child in the manger concerned.

Exclusion Criteria:

* Refusal of parents (lack of consent)
* Refusal of the child according to his ability to understand
* Uninsured social security

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children older than 3 months and less than 6 years kept in nurseries retained, regardless of the duration of custody of the child in the manger concerned.
Sampling Method: Probability Sample
Enrollment: 2001 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Identification of viral shedding | 1 day
  Saliva using small sponges, non-invasive for the viral genome, isolating virus strains and measurement of antibody IgG and IgA.

SECONDARY OUTCOMES:
Evaluate the distribution of different genotypes of strains of CMV | 1 day
  distribution by genotype strains found

CONTACTS AND LOCATIONS:
Overall Officials: Sophie ALAIN, MD, Principal Investigator — Limoges UH
Locations (1):
- Bacteriology, Limoges, France

REFERENCES:
- [Derived] Alain S, Garnier-Geoffroy F, Labrunie A, Montane A, Marin B, Gatet M, Grosjean J, Dufour V, Saugeras M, Postil D, Hantz S. Cytomegalovirus (CMV) Shedding in French Day-Care Centers: A Nationwide Study of Epidemiology, Risk Factors, Centers' Practices, and Parents' Awareness of CMV. J Pediatric Infect Dis Soc. 2020 Dec 31;9(6):686-694. doi: 10.1093/jpids/piz097. PMID 32068854